CLINICAL TRIAL: NCT01421446
Title: Reliability and Validity of Umea Computerized Neuropsychological Battery
Brief Title: Study to Validate a Computerized Neuropsychological Test Battery
Status: Terminated | Type: Observational
Why Stopped: Insufficient subject recruitment
Sponsor: LifeBridge Health (Other)
Responsible Party: Principal Investigator, Michael Williams, Medical Director, Sandra and Malcolm Berman Brain & Spine Institute, LifeBridge Health
Other Study IDs: BSI-LBH 1735
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Elderly
Keywords: Neuropsychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is comparing a new computer-based method of administering neuropsychological tests to the standard method of verbal and paper/pencil tests administered in person by an examiner. The purpose of the research is to determine if the computerized and standard testing methods are equivalent.

DETAILED DESCRIPTION:
Cognitive decline is one of the primary symptom triad of Normal Pressure Hydrocephalus (NPH). Neuropsychological measures have been demonstrated as being effective in the diagnosis of NPH, and in assessing the efficacy of treatment intervention. Hence, neuropsychological assessment is a critical component in the assessment for the presence of NPH. Specifically, measures of attention/concentration, fine motor skills, executive functioning abilities, speed of processing and memory have been found to be useful in the assessment of NPH and treatments thereof.

Neuropsychologists are typically found in large hospitals, academic centers and in urban locations. Neuropsychologists are under represented in rural or low population centers. At the present time, cognitive assessment is frequently limited to a Mini Mental Status Examination. Furthermore, neuropsychological testing can be very expensive for patients, given insurance constraints. Finally, there is no standardized test battery that is used in different centers treating this patient population. The creation of a standard battery that could be used in other NPH centers would promote research collaboration.

A computerized neuropsychological test battery was developed in Umea, Sweden with the specific goal of using tests that are considered to be sensitive to the cognitive profile observed in NPH. The battery was developed in JAVA and Adobe Flash making it platform independent (Runs on Mac, Windows and Linux). The test battery is administered on a touch screen display, where the tests are presented through animations with audio instructions. Before the real test trails are administered, subjects are given practice trials with auditory and visual feedback. For the American version of the test, the auditory stimuli have been translated and recorded in English.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80

Exclusion Criteria:

* Neurological disorder that results in motor or cognitive dysfunction
* Perceptual or motor difficulties that would prevent subjects from taking the assessment
* MMSE score <20
* MoCA score <26
* MAS score >9
* Significant abnormal neurologic examination findings

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy elderly subjects without significant neurologic, psychiatric, cardiovascular, or other systemic disease that impairs neurologic function or cognitive function
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Computer Hydrocephalus Neuropsychological Assessment Versions 1 & 2 | Within 2-5 weeks of enrollment
Standard Hydrocephalus Neuropsychological Assessment: Versions 1 & 2 | Within 2-5 weeks of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Williams, MD, Principal Investigator — LifeBridge Health
Locations (1):
- Sandra and Malcolm Berman Brain & Spine Institute, Baltimore, Maryland, United States